CLINICAL TRIAL: NCT06153667
Title: Prospective, Multi-Center Study Using Bearing nsPVA Embolization Particles for the Treatment of uTErine fibRoids With Uterine Artery Embolization
Brief Title: Bearing nsPVA Embolization for Uterine Artery Embolization (BETTER-UAE)
Acronym: BETTER-UAE
Status: Recruiting | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: UFE-P4-23-01
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bearing nsPVA — Bearing nsPVA Embolization Particles are irregularly-shaped, biocompatible, hydrophilic, nonresorbable particles produced from polyvinyl alcohol. These embolization particles are intended to provide vascular occlusion or reduction of blood flow within target vessels upon selective placement through a variety of catheters. Bearing nsPVA Embolization Particles are used for the embolization of symptomatic (leiomyoma uteri) uterine fibroids.

SUMMARY:
This is a prospective, multicenter, observational, post-market clinical follow-up study in subjects treated with Bearing nsPVA Embolization Particles for uterine fibroid embolization. Data collection will include safety and performance outcome relating to the use of Bearing nsPVA, through 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥ 18 years old at the time of enrollment.
* Subject has symptomatic uterine fibroid(s), suitable to embolization.
* Subject provides written informed consent.

Exclusion Criteria:

* Subject is pregnant.
* Subject has suspected pelvic inflammatory disease or any other pelvic infection.
* Subject has any malignancy of the pelvic region, (e.g., endometrial neoplasia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women ≥ 18 years with symptomatic uterine fibroid(s).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 30 days
  The primary safety endpoint will be the absence of serious device-related adverse events (AEs) through 30 days.
Primary Effectiveness | 6 months
  The primary effectiveness endpoint will be clinical success defined as ≥ 50% improvement in the Uterine Fibroid Symptom and Quality of Life (UFS-QoL) Symptom Severity subscale at 6 months as compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The Alfred Health, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No